CLINICAL TRIAL: NCT04997057
Title: Effect of a Mixture of Probiotics (Lactibiane Reference) in Patients With Irritable Bowel Syndrome Predominantly Constipation and Assessment of a Potential Biomarker (Resolvin D1): an Exploratory Study
Brief Title: A Multistrain Probiotic in Patients With Irritable Bowel Syndrome With Predominant Constipation
Acronym: EPORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: PiLeJe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1674
Record Dates: First submitted 2021-07-19; First posted 2021-08-09 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-03

CONDITIONS: Irritable Bowel Syndrome With Constipation

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study: post-treatment versus baseline comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotics mixture (Other): Daily supplementation with a mixture of probiotics for 12 weeks
  Interventions: Dietary Supplement: Probiotics mixture

INTERVENTIONS:
Dietary Supplement: Probiotics mixture — 12 weeks of daily supplementation with 1 g of probiotics mixture (4.10exp9 colony forming unit/g) containing:
  * Bifidobacterium longum LA 101
  * Lactobacillus helveticus La 102
  * Lactococcus lactis LA 103
  * Streptococcus thermophilus LA 104

SUMMARY:
Probiotics efficacy is mainly assessed by subjective endpoints such as the FDA responder rate or global relief, which partly explain contradictory results obtained in clinical trials with probiotic bacteria. Objective biomarkers of IBS will allow to measure the efficacy of probiotics. In the case of IBS-C, serum resolvin-D1 appears to be an interesting candidate due to its non-invasive and discriminating character compared to a healthy population. It is, inversely correlated with the severity of symptoms. Resolvin-D1 modulates the duration and intensity of inflammation by regulating the transcription of cytokines, chemokines and their receptors as well as other proteins involved in inflammation. Resolvin D1 could serve as a predictor of probiotic response based on its baseline value.

DETAILED DESCRIPTION:
Resolvin D1 levels will be measured in patients with IBS-C as defined by the Rome IV criteria before 6 and 12 weeks after supplementation with a mixture of probiotics. The progression of IBS-C symptoms will also be assessed throughout the study.

The correlation with resolvin D1 levels and the severity of IBS symptoms will be investigated. The efficacy of the probiotic mixture in relieving the symptoms of IBS-C will be measured and compared based on the levels of resolvin D1.

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome with constipation (IBS-C) according to Rome IV criteria ;
* IBS-SSS between 175-300 in the last 10 days ;
* Have experienced abdominal pain ≥ 40 according to the IBS-SSS questionnaire (abdominal pain item) during the last 10 days ;
* Whose abdominal pain / discomfort has had a significant impact on daily life during the past 10 days (impact ≥2 on a 5-point likert scale (from 0: no impact to 5: extreme impact) ;
* Ability to understand instructions and complete questionnaires Nurstrial APP.
* Affiliate or beneficiary of a social security ;
* Having given their free, informed and written consent.

Exclusion Criteria:

* CPRu > 10 mg/l
* Pregnant or breastfeeding woman, woman planning a pregnancy during the study period ;
* Intolerance or proven food allergy ;
* BMI <18.5 kg / m2 or BMI> 35 kg / m2 ;
* Diagnosis or known history of IBS-D, IBS-M, or unclassified forms of IBS, or other gastrointestinal pathologies ;
* With current first-line IBS-C treatment or second-line treatment ;
* alternative non pharmacological treatment ;
* Drug treatment affecting visceral sensitivity or intestinal transit ;
* dietary modification (exclusion of FODMAPs, prebiotic) or lifestyle ;
* Excessive smoking or drinking ;
* Having or planning bariatric surgery,
* With known pathologies affecting gut function ;
* With a deviant eating behavior,
* Treated with antibiotics in the 3 months preceding inclusion,
* Under legal protection,
* Already included in a clinical trial,
* With severely impaired physical/psychological health may affect study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Change of the severity of IBS-C symptoms | At weeks 0, 4, 8 and 12
  Measured by the composite IBS-SSS (Irritable Bowel Syndrome-Severity Scale Scoring) system, compared to the baseline IBS-SSS value.
  Minimum : 0 (best condition) to maximum (worse condition): 500

SECONDARY OUTCOMES:
Change of the severity of addominal pain | At weeks 4, 8 and 12
  Mesured by the Abdominal pain domain of the IBS-SSS (Irritable Bowel Syndrome-Severity Scale Scoring) score compared to the baseline.
  Minimum (best condition) : 0 to maximum (worse condition): 100
Change of the number of days with abdominal pain | At weeks 4, 8 and 12
  Mesured by the Number of days with abdominal pain domain of the IBS-SSS (Irritable Bowel Syndrome-Severity Scale Scoring) score compared to the baseline.
  Minimum (best condition) : 0 to maximum (worse condition): 100
Change of the severity of abdominal distension (bloating) | At weeks 4, 8 and 12
  Mesured by the bloating-distension domain of the IBS-SSS (Irritable Bowel Syndrome-Severity Scale Scoring) score compared to the baseline.
  Minimum (best condition) : 0 to maximum (worse condition): 100
Change of the satisfaction with bowel habits | At weeks 4, 8 and 12
  Mesured by the satisfaction with bowel habits domain of the IBS-SSS (Irritable Bowel Syndrome-Severity Scale Scoring) score compared to the baseline.
  Minimum (best condition) : 0 to maximum (worse condition): 100
Change of the IBS-related quality of life | At weeks 4, 8 and 12
  Mesured by the IBS related quality of life domain of the IBS-SSS (Irritable Bowel Syndrome-Severity Scale Scoring) score compared to the baseline.
  Minimum (best condition) : 0 to maximum (worse condition): 100
Global assessment of symptoms relief | At weeks 4, 8 and 12
  Measured by the Subject's Global Assessment (SGA) of Relief, compared to the baseline
Change of Resolvin-D1 levels | At weeks 8 and 12
  Blood measurement of resolvin-D1 compared to the baseline
Change of CPRu (C Reactive Protein-ultrasensitive) levels | At weeks 8 and 12
  Blood measurement of C Reactive Protein ultrasensitive compared to the baseline
Change of the intestinal microbiota | At weeks 6 and 12
  Biological parameter : Fecal microbiota measured by 16S rRNA gene sequencing compared to baseline
Change of the stool frequency | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  Patient-reported number of stools using an e-diary, compared to baseline
Change of the stools consistency | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  Patient-reported stools consistency by the Bristol Stool Scale, using an e-diary, compared to baseline
Change of the Quality of Life | At weeks 4, 8 and 12
  Measured by Medical Outcomes Study Short-Form General Health Survey Short Form-12 compared to baseline
Change of number of drugs consumption to alleviate the IBS-C symptoms | At weeks 4, 8 and 12
  Patient-reported drug (laxative, spasmolytics) consumption using an e-diary, compared to baseline
Assessing the relationship between resolvin D1 levels and symptoms severity mesured by IBS-SSS symptoms scores | At week 12
  Regression analysis
Assessing the relationship between baseline resolvin D1 levels and response to the probiotics supplementation measured by the responders rate (outcome 17) | At week 12
  Regression analysis
Assessing the responders rate | At weeks 4, 8 and 12
  Number of patients with a decrease in the weekly average of worst abdominal pain in the past 24 hours score (measured daily) of at least 30 percent compared with baseline weekly average and a stool Frequency Weekly Responder is defined as a patient who experiences an increase of at least one complete stool bowel movement per week from baseline.
Assessing the relationship between baseline microbiota and response to the probiotics supplementation measured by the responders rate (outcome 17) | At week 12
  Regression analysis
Assessing the tolerance of the probiotics mixture | At weeks 6 and 12
  Adverse reactions analysis
Assessing the global improvement | At weeks 4, 8 and 12
  Measured by the patient global impression of improvement
Assessing the satisfaction regarding the mixture of probiotics | At weeks 4, 8 and 12
  Measured by a 5 points Likert scale 0 : worse satisfaction to 5 : better satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: GABRIEL PERLEMUTER, PR, Study Director — Hospital Antoine-Béclère
Locations (1):
- CEN Nutriment, Dijon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No